CLINICAL TRIAL: NCT01959152
Title: Evaluation of Hearing Preservation in Adults With Partial Low-Frequency Hearing Implanted With the HiFocus™ Mid-Scala Electrode
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR0513
Record Dates: First submitted 2013-10-08; First posted 2013-10-09 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-04

CONDITIONS: Hearing Loss; Deafness; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases
Keywords: Cochlear Implant; HiRes™ 90K Advantage implant; Cochlear Implantation; HiFocus™ Mid-Scala electrode; Listening Benefits; Adults; Cochlear Implant Benefit; HiRes Fidelity 120™; Electrical Stimulation
MeSH Terms: conditions — Hearing Loss; Deafness; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HiRes90K™ Advantage Cochlear Implant (Experimental): HiRes90K™ Advantage implant with HiFocus™ Mid-Scala electrode will be implanted in adults with a moderate level of hearing loss in the low frequencies and severe-to-profound hearing loss in the mid-to-high frequencies.
  Interventions: Device: HiRes™ 90K Advantage implant with HiFocus™ Mid-Scala electrode

INTERVENTIONS:
Device: HiRes™ 90K Advantage implant with HiFocus™ Mid-Scala electrode

SUMMARY:
The purpose of this study is to determine the feasibility of preserving low-frequency acoustic hearing in adults with a moderate degree of hearing loss in the low frequencies and severe-to-profound hearing loss in the mid-to-high frequencies who are implanted with the HiRes™ 90K Advantage implant with HiFocus™ Mid-Scala electrode.

ELIGIBILITY:
Inclusion Criteria:

* No previous cochlear implant experience
* 18 years of age or older
* Up to a moderate sensorineural hearing loss in the low-to-mid frequencies (pure tone average ≤ 65 dB HL for 125, 250, 500, and 1000 Hz) and a severe-to-profound sensorineural hearing loss in the high frequencies (pure tone average ≥ 70 dB HL for 2,000, 4,000, and 8,000 Hz) in the ear to be implanted
* Aided monosyllabic word score of 10-50% in the ear to be implanted
* Up to a moderate sensorineural hearing loss in the low-to-mid frequencies (pure tone average ≤ 65 dB HL for 125, 250, 500, and 1000 Hz) and a severe-to-profound sensorineural hearing loss in the high frequencies (pure tone average ≥ 70 dB HL for 2,000, 4,000, and 8,000 Hz) in the contralateral (non-implanted) ear
* English language proficiency
* Willingness to participate in all scheduled procedures outlined in the protocol

Exclusion Criteria:

* Previous inner ear surgery
* Cochlear malformation or obstruction that would preclude full insertion of electrode array
* Presence of additional disabilities that would prevent or interfere with participation in the required study procedures
* Medical or psychological conditions that contraindicate surgery or impact the ability to manage an implanted device or the study-related procedures
* Evidence of central auditory lesion or compromised auditory nerve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Low-frequency unaided acoustic hearing thresholds pre and post implantation with the HiFocus™ Mid-Scala electrode array | One month
  Unaided low-frequency acoustic hearing thresholds (under earphones) in the implanted ear one month after device activation will be compared to baseline (pre-implant) thresholds in the same ear for audiometric frequencies 125-1000Hz. Threshold changes from baseline will be calculated as:
  * Complete preservation of hearing: threshold shift ≤ 15 dB
  * Partial preservation of hearing: threshold shift ≥ 16 dB with measurable thresholds
  * No preservation of hearing: no measurable thresholds at ≤ 80 dB HL

SECONDARY OUTCOMES:
Word recognition in quiet pre and post implantation with the HiFocus™ Mid-Scala electrode array | One month
  Word recognition scores in quiet in the implanted ear one month after device activation compared to pre-implant score with a hearing aid

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Dalhousie University, Department of Surgery, Division of Otolaryngology, Halifax, Nova Scotia
  - The Ottawa Hospital, Parkdale Clinic, Audiology Department, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Department of Otolaryngology - Head and Neck Surgery, Toronto, Ontario